CLINICAL TRIAL: NCT00762515
Title: Clinical Study to Evaluate the Treatment of Gingivitis of Two Toothpastes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2007-GIN-03-RR
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2010-12-14 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque | interventions — Fluorides; Triclosan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): commercially available Fluoride only toothpaste
  Interventions: Drug: Fluoride
- B (Active Comparator): Commercially available triclosan/copolymer/fluoride toothpaste
  Interventions: Drug: Triclosan; Drug: Fluoride

INTERVENTIONS:
Drug: Fluoride — Brush teeth two times daily for 6 weeks
  Arms: A
Drug: Triclosan — Brush two times daily for 6 weeks
  Arms: B
Drug: Fluoride — Brush two times daily for 6 weeks
  Arms: B

SUMMARY:
The objective is to compare two commerical oral products for the treatment of gingivitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers 18-65 years of age
2. Good general health
3. Must sign informed consent form
4. Minimum of 16 natural uncrowned teeth (excluding third molars) must be present.
5. No history of allergy to personal care consumer products, or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study.
6. Dental Selection Criteria: Gingivitis patients with a minimum of 16 gradable teeth with a minimum of 6 sites with a GI score of ≥ 3. Subjects will be stratified according to gingivitis severity. Average full mouth GI score should be in the range of 2.0 - 2.5. heavy plaque formers should be avoided. Target a full mouth PI (Quigley-Hein) to be in the range of 1.5-3.0

Exclusion Criteria:

1. Subjects unable or unwilling to sign the informed consent form.
2. Medical condition which requires pre-medication prior to dental visits/procedures
3. Moderate or advanced periodontal disease
4. History of allergy to iodine
5. History of thyroid disease
6. History of diabetes
7. 2 or more decayed untreated dental sites at screening.
8. Other disease of the hard or soft oral tissues.
9. Impaired salivary function (e.g. Sjogren's syndrome or head and neck irradiation).
10. Use of medications that are currently affect salivary flow.
11. Use of antibiotics or antimicrobial drugs within 30 days prior to study visit #1.
12. Pregnant or nursing women.
13. Participation in any other clinical study within 1 week prior to enrollment into this study.
14. Use of tobacco products
15. Subjects who must receive dental treatment during the study dates.
16. Current use of Antibiotics for any purpose.
17. Presence of an orthodontic appliance.
18. History of allergy to common dentifrice ingredients
19. Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)
20. Women of childbearing potential and not on birth control (Diaphragm, birth control pills or implants, IUD (Intrauterine device), condoms).
21. Smoker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Kinane, BDS, Principal Investigator
Locations (1):
- University of Louisville, School of Dentistry, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects recruited by the PI at the clinical site.
Pre-assignment Details: Screening for subjects that met the overall oral health criteria. Followed by a 1 week washout prior to starting any study treatments or procedures.
Groups:
- A -Placebo Comparator: Fluoride toothpaste
- B- Active Comparator: Fluoride/triclosan toothpaste (Total)
Period: Overall Study
Arm/Group | A -Placebo Comparator | B- Active Comparator
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A -Placebo Comparator | B- Active Comparator | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Control Established Plaque in Adults
Description: Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth. Total Plaque score=sum of all scores divided by the number of sites (teeth) scored.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | A -Placebo Comparator | B- Active Comparator
Number analyzed (Participants) | 22 | 22
Units on a scale | 2.42 (0.47) | 2.45 (0.53)
Statistical Analysis 1: Comparison: A -Placebo Comparator vs B- Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, ANCOVA; baseline is used a factor

2. Secondary Outcome: Control Gingivitis in Adults
Description: Gingivitis Index (GI) is described as Units on a scale 0 to 3 (0 = no inflammation,1 = Mild inflammation - slight change in color and little change in texture 2 = Moderate inflammation - moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding. GI score = Sum of all scores divided by the number of sites (teeth scored).
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | A -Placebo Comparator | B- Active Comparator
Number analyzed (Participants) | 22 | 22
Units on a scale | 0.54 (0.16) | 0.63 (0.19)
Statistical Analysis 1: Comparison: A -Placebo Comparator vs B- Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, ANCOVA; baseline to be used a factor

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | A -Placebo Comparator | B- Active Comparator
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less